CLINICAL TRIAL: NCT00294385
Title: A Randomized Phase III Study Comparing Concomitant Docetaxel Plus Gemcitabine to Sequential Therapy of Docetaxel Followed by Gemcitabine in Anthracycline-Pretreated Metastatic or Locally Recurrent Breast Cancer Patients
Brief Title: Study Comparing Concomitant Docetaxel + Gemcitabine to Sequential Therapy of Docetaxel Followed by Gemcitabine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Central European Cooperative Oncology Group (Other)
Responsible Party: Prof. Dr. Thomas Brodowicz, CECOG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CECOG/BC 1.3.002
Record Dates: First submitted 2006-02-20; First posted 2006-02-22 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Docetaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemcitabine, Docetaxel (Active Comparator): Arm A (concomitant arm), Gemcitabine 1000 mglm2 will be administered intravenously on Days 1 and 8, repeated on Day 22. Docetaxel 75 mg/m2 will be given on Day 8 (before Gemcitabine), repeated on Day 22. This 3-week schedule defines a cycle of treatment for this arm. Overall 8 cycles will be administered.
  Interventions: Drug: Docetaxel; Drug: Gemcitabine, Docetaxel
- Docetaxel (Active Comparator): Arm B (sequential arm) four cycles of Docetaxel 100 mg/m2 an Day 1, repeated an Day 22, followed by four cycles of Gemcitabine 1250 mg/m2 an a Day 1 and 8, repeated an Day 22, will be given. Both drugs will be administered in a 3-week schedule.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel
Drug: Gemcitabine, Docetaxel — Arm A (concomitant arm), Gemcitabine 1000 mglm2 will be administered intravenously on Days 1 and 8, repeated on Day 22. Docetaxel 75 mg/m2 will be given on Day 8 (before Gemcitabine), repeated on Day 22. This 3-week schedule defines a cycle of treatment for this arm. Overall 8 cycles will be administered.
  Arms: Gemcitabine, Docetaxel
Drug: Docetaxel — rm B (sequential arm) four cycles of Docetaxel 100 mg/m2 an Day 1, repeated an Day 22, followed by four cycles of Gemcitabine 1250 mg/m2 an a Day 1 and 8, repeated an Day 22, will be given. Both drugs will be administered in a 3-week schedule.
  Arms: Docetaxel

SUMMARY:
The purpose of this study is to compare the Time To Disease Progression (TTDP) between those patients with unresectable, locally recurrent or metastatic breast cancer who are treated with concomitant Docetaxel plus Gemcitabine to those patients treated with sequential therapy of Docetaxel followed by Gemcitabine.

DETAILED DESCRIPTION:
This is an open, multicenter, two-armed Phase III study

Patients will be randomized to either of the following two arms:

Arm A (concomitant arm), Gemcitabine 1000 mglm2 will be administered intravenously on Days 1 and 8, repeated on Day 22. Docetaxel 75 mg/m2 will be given on Day 8 (before Gemcitabine), repeated on Day 22. This 3-week schedule defines a cycle of treatment for this arm. Overall 8 cycles will be administered.

Arm B (sequential arm) four cycles of Docetaxel 100 mg/m2 an Day 1, repeated an Day 22, followed by four cycles of Gemcitabine 1250 mg/m2 an a Day 1 and 8, repeated an Day 22, will be given. Both drugs will be administered in a 3-week schedule.

Bimonthly follow-up for patients without confirmed disease progression until progression of disease. Long-term follow-up for patients with confirmed disease progression will be done in 4 intervals.

For therapy control frequent blood chemistry and hematology, physical examination, weight control, potential adverse events and imaging procedures (CT, X-ray, MRI, Bone scan) am foreseen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic or cytologic diagnosis of breast cancer with evidence of unresectable, locally recurrent, or metastatic disease.
* Females, 18 to 75 years of age
* pre-treated with ONE anthracyclines containing chemotherapy either in neoadjuvant/adjuvant or 1st line metastatic setting will be enrolled into the study
* Patients with clinically measurable lesions will be enrolled in this study. Measurability is determined according to RECIST criteria
* Performance status of 70 or higher on the Karnofsky Performance Scale
* Adequate bone marrow reserve
* Adequate liver function
* Adequate renal function
* Informed consent form patient or guardian
* Childbearing potential either terminated by surgery, radiation, or menopause, use of an approved contraceptive method

Exclusion Criteria:

* Active infection (at the discretion of the investigator).
* Known or suspected brain metastases requiring steroid or radiation treatment.
* Pregnancy (recent negative urine pregnancy test for pre-menopausal patients mandatory)
* Breast-feeding
* Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator).
* Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin).
* Bone metastases, pleural effusion, or ascites as the only site of disease.
* Bone marrow transplantation or autologous stern cell infusion following high-dose chemotherapy for adjuvant or metastatic disease.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2002-06; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
to compare the Time To Disease Progression between those patients with unresectable, locally recurrent or metastatic breast cancer who are treated with concomitant Docetaxel plus Gemcitabine to those patients treated with sequential therapy of Doc

SECONDARY OUTCOMES:
Overall response rate
Response duration
Overall survival
Characterize changes in performance status, patient-reported pain, and disease-related symptoms in each arm
Characterize the nature of the toxicities experienced in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Wiltschke, Prof, Principal Investigator — Univ. Klinik f. Innere Medizin I
Locations (17):
- Austria (3):
  - 2. Med. Abteilung - LKH-Steyr, Steyr
  - Hanusch KrankenhausHämatologisch-Onkologisches Zentrum, Vienna
  - Intere IV Krankenhaus Wels, Wels
- Bulgaria (2):
  - Cancer Center Plovdiv, Plovdiv
  - SBALO National Oncology Center, Sofia
- Czechia (5):
  - FN U sv. Anny, Brno
  - Nemocnice Ceske Budejovice, Ceske
  - FN Hradec Kralove, Hradec Králové
  - FN Bulovka, Prague
  - Charles University Prague, Dep of Oncology, Prague
- Israel (3):
  - Rambam Medical Center, Oncol. Dep, Haifa
  - Tel Aviv Sourasky Medical Center, Div of Oncology, Tel Aviv
  - "Sheba" Medical Center, Dep of Oncology, Tel Litwinsky
- Lebanon (2):
  - American University of Beirut, Medical Center, Beirut
  - Rizk Hospital, Beirut
- Klinika Onkologii CMuJ, Krakow, Poland
- Nomocnica Sv. Alzbety, Narodny Onkologicky Ustav, Bratislava, Slovakia